CLINICAL TRIAL: NCT01642212
Title: Oral Budesonide Suspension (OBS) in Adolescent and Adult Subjects (11-40 Years of Age)With Eosinophilic Esophagitis: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study With an Open Label Extension
Brief Title: OBS in Adolescent and Adults With EOE: A Phase II, Randomized, Double-Blind, Placebo Controlled, Study With an Open Label Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPI-101-06
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Budesonide Suspension (Experimental): Taken once or twice daily for up to 40 weeks
  Interventions: Drug: Oral Budesonide Suspension (MB-9)
- Matching Placebo (Placebo Comparator): Taken once or twice daily for 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Budesonide Suspension (MB-9) — OBS suspension to be taken bid over a 16 week course of double blind therapy and OBS suspension to be taken qd to bid during a 24 week optional open label extension period
  Arms: Oral Budesonide Suspension
Drug: Placebo
  Arms: Matching Placebo

SUMMARY:
This is a clinical trial to test an experimental drug for the treatment of Eosinophilic Esophagitis (EoE)

DETAILED DESCRIPTION:
Eosinophilic Esophagitis (EoE) is an inflammatory disorder of the esophagus and is a recognized clinical entity. Symptoms include feeding problems, heartburn, regurgitation, vomiting, abdominal pain and food impaction. The symptoms of EoE may be similar to gastroesophageal reflux disease (GERD) but do not resolve with gastric acid suppression. EoE is defined histologically as the presence of > 15 intraepithelial eosinophils per high power fields on one or more esophageal biopsy specimens.

This Phase II study is comparing oral budesonide (OBS) to placebo to demonstrate that OBS induces a histologic response and a symptom response using a Dysphagia Symptom Questionnaire over a 16 week course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, age 11-40
* Histologic evidence of EoE
* History of clinical symptoms of EoE including dysphagia
* Willing to continue with dietary, environmental or medical therapy
* Ability to read and understand english
* Written Consent

Exclusion Criteria:

* Any Medical condition that may compromise the safety of the subjects or interfere with the signs and symptoms of EoE
* Use of immunomodulatory therapy
* Current use of swallowed corticosteroids
* Esophageal strictures,varices or upper GI bleed
* Other current diseases of the GI tract
* Current viral infection or immunodeficiency condition
* Pregnancy
* Hypersensitivity to budesonide
* History of non compliance

Ages: 11 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2014-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (23):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - UCSD Rady Children's Hospital, San Diego, California
  - The Children's Hospital, Aurora, Colorado
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Northwestern Scool of Medicine, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Center for Children's Digestive Health, Park Ridge, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - The Mayo Clinic, Rochester, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Cincinnati Center for Eosinophilic Disorders, Cincinnati, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Children's Center for Digestive Health, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah Healthcare, Salt Lake City, Utah
  - Carilion Pediatric Gastroenterology, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mukkada VA, Gupta SK, Gold BD, Dellon ES, Collins MH, Katzka DA, Falk GW, Williams J, Zhang W, Boules M, Hirano I, Desai NK. Pooled Phase 2 and 3 Efficacy and Safety Data on Budesonide Oral Suspension in Adolescents with Eosinophilic Esophagitis. J Pediatr Gastroenterol Nutr. 2023 Dec 1;77(6):760-768. doi: 10.1097/MPG.0000000000003948. Epub 2023 Sep 18. PMID 37718471
- [Derived] Dellon ES, Collins MH, Katzka DA, Hudgens S, Lan L, Williams J, Vera-Llonch M, Hirano I. Improvements in Dysphagia and Pain With Swallowing in Patients With Eosinophilic Esophagitis Receiving Budesonide Oral Suspension. Clin Gastroenterol Hepatol. 2021 Apr;19(4):699-706.e4. doi: 10.1016/j.cgh.2020.03.060. Epub 2020 Apr 6. PMID 32272243
- [Derived] Hirano I, Dellon ES, Collins MH, Williams J, Lan L, Katzka DA. Clinical Features at Baseline Cannot Predict Symptom Response to Placebo in Patients With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2126-2128.e1. doi: 10.1016/j.cgh.2018.11.045. Epub 2018 Nov 28. PMID 30502508
- [Derived] Dellon ES, Katzka DA, Collins MH, Gupta SK, Lan L, Williams J, Hirano I. Safety and Efficacy of Budesonide Oral Suspension Maintenance Therapy in Patients With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2019 Mar;17(4):666-673.e8. doi: 10.1016/j.cgh.2018.05.051. Epub 2018 Jun 12. PMID 29902649
- [Derived] Dellon ES, Katzka DA, Collins MH, Hamdani M, Gupta SK, Hirano I; MP-101-06 Investigators. Budesonide Oral Suspension Improves Symptomatic, Endoscopic, and Histologic Parameters Compared With Placebo in Patients With Eosinophilic Esophagitis. Gastroenterology. 2017 Mar;152(4):776-786.e5. doi: 10.1053/j.gastro.2016.11.021. Epub 2016 Nov 23. PMID 27889574

RESULTS

PARTICIPANT FLOW:
Groups:
- Single-blind Placebo: Eligible participants entered a 4-week, single-blind, placebo baseline period. Participants ingested the first dose of placebo in the clinic in the presence of study center personnel, and the remaining doses were ingested at home. Participants took placebo twice daily (bid); once in the morning after breakfast and once in the evening at bedtime; the volume per dose was 10 mL of oral liquid.
- Double-blind Placebo: Participants took placebo twice daily (bid) at home for 12 weeks. Study drug was administered once in the morning after breakfast and once in the evening at bedtime; the volume per dose was 10 mL of oral liquid.
- Double-blind Oral Budesonide Suspension (OBS) 2 mg: Participants took 2 mg OBS (formulation MB-9) twice daily (bid) at home for 12 weeks. Study drug was administered once in the morning after breakfast and once in the evening at bedtime; the volume per dose was 10 mL of oral liquid.
- Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg; Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg: During the first 12 weeks of open-label extension treatment, participants took 2 mg OBS (formulation MB-9) once daily (qd) at bedtime. The volume per dose was 10 mL of oral liquid (10 mL qd; 0.2 mg/mL). Thereafter, an optional dose increase to 1.5 mg twice daily (bid) (7.5 mL bid; 0.2 mg/mL) and then to 2 mg bid (10 mL bid; 0.2 mg/mL) was allowed for subjects whose response to the 2 mg once daily dose was inadequate, as determined by the Investigator; a dose decrease to 2 mg once daily was allowed at any time.
Period: Single-blind Baseline
Arm/Group | Single-blind Placebo | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg | Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg | Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg
Started | 119 | 0 | 0 | 0 | 0
Completed | 93 | 0 | 0 | 0 | 0
Not Completed | 26 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Eligibility Criteria | 26 | 0 | 0 | 0 | 0
Period: Double-blind Treatment
Arm/Group | Single-blind Placebo | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg | Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg | Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg
Started | 0 | 42 | 51 | 0 | 0
Completed | 0 | 39 | 49 | 0 | 0
Not Completed | 0 | 3 | 2 | 0 | 0
Not completed — Other | 0 | 2 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Period: Open-label Extension
Arm/Group | Single-blind Placebo | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg | Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg | Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg
Started | 0 | 0 | 0 | 37 (Two participants completed double-blind treatment but did not enter the open-label extension.) | 45 (Four participants completed double-blind treatment but did not enter the open-label extension.)
Completed | 0 | 0 | 0 | 27 | 37
Not Completed | 0 | 0 | 0 | 10 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 7 | 4
Not completed — Consent Withdrawn | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set, defined as all randomized participants who received at least 1 dose of double-blind study drug (placebo or OBS); subjects were analyzed based on the actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg | Total
Number analyzed (Participants) | 42 | 51 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (7.50) | 22.3 (7.92) | 21.6 (7.73)
Age, Customized [Count of Participants; unit: Participants]
  <18 Years Of Age | 17 | 18 | 35
  >/= 18 Years Of Age | 25 | 33 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 29 | 35 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Were Histologic Responders
Description: Histologic response was defined as a peak eosinophil count </= 6/high power field (light microscopy) (HPF) across all esophageal levels at the final treatment evaluation (Week 16). An independent, central pathologist determined the peak eosinophil count from the proximal, mid-, and distal levels and selected the maximum peak value. Histopathology data were collected in a blinded fashion.
Time Frame: Week 16
Population: The modified Intent-to-Treat (MITT) Analysis Set: all randomized participants who received at least 1 dose of double-blind study drug and had both an evaluable post-baseline biopsy during the treatment period and a post-baseline DSQ score. Participants were analyzed based on the randomization schedule, regardless of the treatment actually received.
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants | 2.6 | 38.8
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Primary Outcome: Change From Baseline in The Dysphagia Symptom Questionnaire (DSQ) Score at The Final Treatment Period Evaluation
Description: Participants' dysphagia symptoms were evaluated using the 4-item DSQ. The questionnaire was developed by the Sponsor, as an ePRO measure, according to the principles of the Final Guidance for Industry for Patient Reported Outcome Measures (PRO Guidance December 2009). All participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing).The DSQ score was calculated based on responses to Questions 2 and 3 [14 x (sum of points from Questions 2 and 3 in the daily DSQ)/number of diaries with non-missing data]. Baseline was the DSQ score of the 14-day period before randomization. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, Week 16
Population: The MITT Analysis Set: all randomized participants who received at least 1 dose of double-blind study drug and had both an evaluable post-baseline biopsy during the treatment period and a post-baseline DSQ score. Participants were analyzed based on the randomization schedule, regardless of the treatment actually received.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale | -7.53 (1.910) | -14.27 (1.682)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Test type: Superiority or Other; p = 0.0096, ANCOVA — LS mean estimates were determined using an ANCOVA model including treatment group as a factor and the baseline score as a covariate; LS mean difference = -6.75, 95% CI 2-sided [-11.808 to -1.687]

3. Secondary Outcome: Change From Baseline in The DSQ Score Over Time
Description: as for outcome 2
Time Frame: Baseline, Weeks 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale
  Week 8, n = 37, 49 | -4.92 (1.673) | -7.41 (1.453)
  Week 12, n = 36, 49 | -7.42 (2.065) | -10.33 (1.770)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 8; Test type: Superiority or Other; p = 0.2649, ANCOVA — LS mean estimates were determined using the ANCOVA model including treatment group as a factor and baseline DSQ score as a covariate; LS mean difference = -2.49, 95% CI 2-sided [-6.895 to 1.920]
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 12; Test type: Superiority or Other; p = 0.2878, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -2.91, 95% CI 2-sided [-8.322 to 2.501]

4. Secondary Outcome: Change From Baseline in The DSQ Score For The 50th Percentile of Participants at The Final Treatment Period Evaluation
Description: A cumulative distribution function curve was constructed to illustrate the cumulative proportion of participants (x-axis) vs. the change in the DSQ score from baseline to the final treatment evaluation (y-axis). The 50th percentile is participants with a DSQ score that is in the middle of the distribution of all scores. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale | -6.35 | -11.20

5. Secondary Outcome: Percent of Participants With a Peak Eosinophil Count </= 15/High Power Field (Light Microscopy) (HPF) And </= 1/HPF at The Final Treatment Period Evaluation
Description: An independent, central pathologist determined the peak eosinophil count from the proximal, mid-, and distal levels and selected the maximum peak value across all available esophagus levels. Histopathology data were collected in a blinded fashion. The values reported are for participants with histologic response.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  </= 15 Eosinophils/HPF | 7.9 | 46.9
  </= 1 Eosinophils/HPF | 0 | 30.6
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of </= 15 Eosinophils/HPF; Test type: Superiority or Other; p = 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of </= 1 Eosinophils/HPF; Test type: Superiority or Other; p < 0.0001, Fisher Exact

6. Secondary Outcome: Percent of Participants With a >/= 30% And >/= 50% Reduction In The DSQ Score From Baseline to The Final Treatment Period Evaluation
Description: Participants' dysphagia symptoms were evaluated using the 4-item DSQ. The questionnaire was developed by the Sponsor, as an ePRO measure, according to the principles of the Final Guidance for Industry for Patient Reported Outcome Measures (PRO Guidance December 2009). All participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing).The DSQ score was calculated based on responses to Questions 2 and 3 [14 x (sum of points from Questions 2 and 3 in the daily DSQ)/number of diaries with non-missing data]. Baseline was the DSQ score of the 14-day period before randomization.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  >/= 30% DSQ Score Reduction | 44.7 | 69.4
  >/= 50% DSQ Score Reduction | 39.5 | 63.3
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of >/= 30% DSQ score reduction; Test type: Superiority or Other; p = 0.0206, Pearson's chi-square
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of >/= 50% DSQ score reduction; Test type: Superiority or Other; p = 0.0275, Pearson's chi-square

7. Secondary Outcome: Percent of Participants Who Were Overall Responders at The Final Treatment Period Evaluation
Description: Overall response was defined as a reduction in the 2-week DSQ score of >/= 30% and >/= 50% from baseline to the final treatment period evaluation and a peak eosinophil count of </= 6/high power field (light microscopy) (HPF) across all available esophageal levels at the final treatment period evaluation. An independent, central pathologist determined the peak eosinophil count from the proximal, mid-, and distal levels and selected the maximum peak value. Histopathology data were collected in a blinded fashion.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  Responder and >/= 30% DSQ Score Reduction | 2.6 | 26.5
  Responder and >/= 50% DSQ Score Reduction | 2.6 | 20.4
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of response and >/= 30% DSQ score reduction; Test type: Superiority or Other; p = 0.0026, Fisher Exact
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of response and >/= 50% DSQ score reduction; Test type: Superiority or Other; p = 0.0199, Fisher Exact

8. Secondary Outcome: Change From Baseline in The Histopathologic Epithelial Features Combined Total Score at The Final Treatment Period Evaluation
Description: Each esophageal biopsy specimen was evaluated microscopically by an independent, central pathologist for signs of epithelial inflammation and lamina propria fibrosis. Histopathologic epithelial features of each available esophageal level biopsy consisting of basal layer hyperplasia, eosinophil peak, dilated intercellular spaces, eosinophil microabcesses, surface layering, surface alteration, and apoptotic epithelial cells were scored and summed. Histopathology data were collected in a blinded fashion. Histopathology epithelial features were scored for both grade and stage. Each feature had a possible score of 0-3 for grade as well as stage. Thus each of the 3 levels had a possible score of 21, and a possible total grade or stage score of 63 for a maximum combined score of 126. The grade and stage score of the lamina propria was not included because the biopsy material was not available. A negative change from baseline indicates that epithelial inflammation decreased.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale | -1.41 (2.970) | -23.75 (2.602)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean based on the ANCOVA model including treatment group as a factor and baseline as a covariate; LS mean difference = -22.34, 95% CI 2-sided [-30.345 to -14.334]

9. Secondary Outcome: Change From Baseline in The Total Endoscopy Score at The Final Treatment Period Evaluation
Description: The gross endoscopic appearance of the esophageal surface was evaluated by a blinded study center physician. Endoscopic findings with separate evaluations of the proximal and distal esophagus were recorded with respect to 5 major categories, including exudates or plaques, fixed esophageal rings, edema, furrows, and strictures. The endoscopy score was the sum of the scores for the 5 major categories - grade 0-1 for strictures; grade 0-2 for exudates or plaques, edema, and furrows; and grade 0-3 for fixed esophageal rings for the proximal and distal locations. The maximum endoscopy score was 10 points for each location (proximal and distal), and the total endoscopy score was the sum of the scores for the proximal and distal locations (maximum total score of 20 points). Baseline was defined as the endoscopy score at screening. A negative change from baseline indicates that appearance improved.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale | 0.19 (0.530) | -3.58 (0.466)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — LS mean estimates based on the ANCOVA model including treatment group as a factor and baseline value as a covariate; LS mean difference = -3.76, 95% CI 2-sided [-5.172 to -2.358]

10. Secondary Outcome: Change From Baseline in The Peak Eosinophil Count at Each Available Esophageal Level at The Final Treatment Period Evaluation
Description: An independent, central pathologist determined the peak eosinophil count from the proximal, mid-, and distal levels and selected the maximum peak value across all available esophagus levels. Histopathology data were collected in a blinded fashion. Baseline was defined as the score at screening. A negative change from baseline indicates that eosinophil count decreased.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: eosinophils/HPF
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
eosinophils/HPF
  Proximal, n = 32, 45 | -30.06 (6.798) | -65.56 (5.704)
  Mid-, n = 36, 46 | -17.34 (9.244) | -76.90 (8.173)
  Distal, n = 38, 49 | -1.90 (9.852) | -69.28 (8.667)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of proximal eosinophil count; Test type: Superiority or Other; p = 0.0002, ANCOVA — LS mean estimates based on the ANCOVA model including treatment group as a factor and baseline value as a covariate; LS mean difference = -35.50, 95% CI 2-sided [-53.438 to -17.570]
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of mid- eosinophil count; Test type: Superiority or Other; p < 0.0001, ANCOVA — LS mean estimates based on the ANCOVA model including treatment group as a factor and baseline value as a covariate; LS mean difference = -59.56, 95% CI 2-sided [-84.173 to -34.948]
Statistical Analysis 3: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of distal eosinophil count; Test type: Superiority or Other; p < 0.0001, ANCOVA — LS mean estimates based on the ANCOVA model including treatment group as a factor and baseline value as a covariate; LS mean difference = -67.38, 95% CI 2-sided [-93.573 to -41.180]

11. Secondary Outcome: Change From Baseline in The Physician's Global Assessment (PGA) of Disease Activity at The Final Treatment Period Evaluation
Description: The physician Investigator (or qualified physician's assistant or nurse practitioner) completed the PGA to provide the global assessment of eosinophilic esophagitis (EoE) disease activity using a 0 to 100 mm visual analog scale (VAS) scale. The VAS is a 100 mm horizontal line on which the right extreme (100) is labeled "worst possible disease activity" and the left extreme (0) is labeled "no disease activity". The PGA raters were instructed to consider the line for the VAS a continuum with their own medical opinion or judgment of extremes on either end and to draw a vertical line at a point that best approximates the participant's current level of EoE disease activity. A negative change from baseline indicates that disease activity decreased.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale | -10.16 (4.199) | -28.61 (3.695)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Test type: Superiority or Other; p = 0.0015, ANCOVA — LS mean estimates were based on the ANCOVA model including treatment group as a factor and baseline value as a covariate; LS mean difference = -18.44, 95% CI 2-sided [-29.593 to -7.293]

12. Secondary Outcome: Distribution of Responses For The Patient Global Impression of Change (PGIC) Survey at The Final Treatment Evaluation
Description: Participants evaluated the change in their dysphasia (food passing slowly/difficulty swallowing) since the start of the study (screening) by choosing 1 of 7 responses on the PGIC survey: much worse (-3), worse (-2), a little worse (-1), no change (0), a little better (1), better (2), or much better (3). The values reported are the percent of participants who chose that response.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  Much Worse | 0 | 0
  Worse | 2.6 | 2.1
  A Little Worse | 13.2 | 2.1
  No Change | 15.8 | 12.5
  A Little Better | 28.9 | 25.0
  Better | 28.9 | 25.0
  Much Better | 10.5 | 33.3
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of distribution of scores across all responses; Test type: Superiority or Other; p = 0.1170, Cochran-Mantel-Haenszel — P-value for comparison of the treatment difference was determined by Cochran-Mantel-Haenszel row mean score test

13. Secondary Outcome: Percent of Participants With Improved Symptoms on The Eosinophilic Esophagitis (EoE) Symptom Survey at The Final Treatment Period Evaluation
Description: The EoE survey assessed the following symptoms: heartburn, chest pain, regurgitation, abdominal pain, nausea, and vomiting. Participants indicated, by checking a box, if they had a change in symptoms (excluding dysphasia or food impaction) within the past 2 weeks. Baseline was defined as the assessment before randomization. Responses were as follows regarding symptoms at the final treatment evaluation: Improved - participant reported a specific symptom at baseline, but changed to no specific symptom ('Yes' to 'No'); No change - participant reported or did not report a specific symptom at both baseline and the final treatment evaluation; Worsened -participant did not report a specific symptom at baseline, but changed to report that specific symptom ('No' to 'Yes').
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  Heartburn | 10.5 | 18.4
  Chest Pain | 23.7 | 18.4
  Regurgitation | 15.8 | 20.4
  Abdominal Pain | 15.8 | 10.2
  Nausea | 10.5 | 16.3
  Vomiting | 5.3 | 4.1
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of heartburn; Test type: Superiority or Other; p = 0.1947, Cochran-Mantel-Haenszel — P-value for comparison of the treatment difference at baseline vs. final treatment evaluation was determined by a Cochran-Mantel-Haenszel row mean score test. All responses (improved, no change, worsened) were analyzed collectively for each symptom
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of chest pain; Test type: Superiority or Other; p = 0.8029, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of regurgitation; Test type: Superiority or Other; p = 0.4963, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of abdominal pain; Test type: Superiority or Other; p = 0.5257, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of nausea; Test type: Superiority or Other; p = 0.5219, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of vomiting; Test type: Superiority or Other; p = 0.2886, Cochran-Mantel-Haenszel — [p-value comment as in outcome 13, analysis 1]

14. Secondary Outcome: Percent of Participants With No Change in Symptoms on The EoE Symptom Survey at The Final Treatment Period Evaluation
Description: as for outcome 13
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  Heartburn | 86.8 | 71.4
  Chest Pain | 68.4 | 71.4
  Regurgitation | 71.1 | 73.5
  Abdominal Pain | 76.3 | 85.7
  Nausea | 86.8 | 77.6
  Vomiting | 81.6 | 91.8

15. Secondary Outcome: Percent of Participants With Worsened Symptoms on The EoE Symptom Survey at The Final Treatment Period Evaluation
Description: as for outcome 13
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  Heartburn | 2.6 | 10.2
  Chest Pain | 7.9 | 10.2
  Regurgitation | 13.2 | 6.1
  Abdominal Pain | 7.9 | 4.1
  Nausea | 2.6 | 6.1
  Vomiting | 13.2 | 4.1

16. Secondary Outcome: Percent of Participants Without Symptoms on The EoE Symptom Survey at The Final Treatment Period Evaluation
Description: This outcome assessed the symptoms of participants who were symptom-free at baseline. The EoE survey assessed the following symptoms: heartburn, chest pain, regurgitation, abdominal pain, nausea, and vomiting. Participants indicated, by checking a box, if they had a change in symptoms (excluding dysphasia or food impaction) within the past 2 weeks. Baseline was defined as the assessment before randomization. Responses were as follows regarding symptoms at the final treatment evaluation: No change - participant did not report a specific symptom at both baseline and the final treatment evaluation; Worsened -participant did not report any symptom at baseline, but changed to report at least 1 symptom at the final treatment evaluation.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants | 71.1 | 83.7
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of symptoms of participants with no symptoms at baseline; Test type: Superiority or Other; p = 0.1600, Cochran-Mantel-Haenszel — P-value for comparison of the treatment difference at baseline vs. final treatment evaluation was determined by a Cochran-Mantel-Haenszel row mean score test. Both responses (no change, worsened) were analyzed collectively

17. Secondary Outcome: Percent of Participants With New Symptoms on The EoE Symptom Survey at The Final Treatment Period Evaluation
Description: This outcome assessed the symptoms of participants who were symptom-free at baseline. The EoE survey assessed the following symptoms: heartburn, chest pain, regurgitation, abdominal pain, nausea, and vomiting. Participants indicated, by checking a box, if they had a change in symptoms (excluding dysphasia or food impaction) within the past 2 weeks. Baseline was defined as the assessment before randomization. Responses were as follows regarding symptoms at the final treatment evaluation: No change - participant reported or did not report a specific symptom at both baseline and the final treatment evaluation; Worsened -participant did not report any symptom at baseline, but changed to report at least 1 symptom at the final treatment evaluation.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants | 28.9 | 16.3

18. Secondary Outcome: Percent of Participants Who Were Symptom Responders on The DSQ+Pain Scale at The Final Treatment Period Evaluation
Description: Participants' dysphagia symptoms were evaluated using the 4-item DSQ. The questionnaire was developed by the Sponsor, as an ePRO measure, according to the principles of the Final Guidance for Industry for Patient Reported Outcome Measures (PRO Guidance December 2009). All participants used a diary, and responded to Question 1 (did you eat solid food) and Question 2 (did food pass slowly or get stuck). If the answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Question 3 (did you have to do anything to make the food go down or get relief) and Question 4 (extent to which the participant experienced pain while swallowing).The DSQ+pain response was defined as a >/= 30% and >/= 50% reduction from baseline in the combined score from Questions 2, 3, and 4. The 2-week DSQ+pain score was calculated by adding points from Questions 2, 3, and 4 and then taking the average of the available scores over each 2-week interval.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percent of participants
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percent of participants
  >/= 30% DSQ+pain Score Reduction | 47.4 | 67.3
  >/= 50% DSQ+pain Score Reduction | 39.5 | 65.3
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of >/= 30% DSQ+pain score reduction; Test type: Superiority or Other; p = 0.0606, Pearson's chi-square
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of >/= 50% DSQ+pain score reduction; Test type: Superiority or Other; p = 0.0165, Pearson's chi-square

19. Secondary Outcome: Percent of Days That Participants Reported That They Avoided Solid Food During The Baseline And Treatment Periods
Description: Participants' dysphagia symptoms were evaluated using the 4-item DSQ. The questionnaire was developed by the Sponsor, as an ePRO measure, according to the principles of the Final Guidance for Industry for Patient Reported Outcome Measures (PRO Guidance December 2009). All participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). Values were calculated for all the days that Question 1 was answered from 14 days prior to baseline visit up to the final treatment period evaluation.
Time Frame: From 14 days prior to the baseline visit to the final treatment period evaluation
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: percentage of days
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
percentage of days | 1.2 [0.0 to 1.1] | 0.7 [0.0 to 1.2]
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Test type: Superiority or Other; p = 0.7817, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in The Scores of DSQ Question 1 During The Treatment Period
Description: Participants' dysphagia symptoms were evaluated using the 4-item DSQ. The questionnaire was developed by the Sponsor, as an ePRO measure, according to the principles of the Final Guidance for Industry for Patient Reported Outcome Measures (PRO Guidance December 2009). All participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). Question 1 is rated as Yes (score=0) or No (score=1); higher values indicate a worse outcome. Baseline was the DSQ score of the 14-day period before randomization. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, Weeks 8, 12, and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale
  Week 8, n = 37, 49 | 0.02 (0.050) | -0.08 (0.043)
  Week 12, n = 36, 49 | 0.05 (0.091) | 0.02 (0.078)
  Week 16, n = 38, 49 | 0.05 (0.079) | 0.06 (0.069)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 8; Test type: Superiority or Other; p = 0.1686, ANCOVA — Estimates are determined using an ANCOVA model including treatment group as a factor and baseline DSQ score as a covariate; LS mean difference = -0.09, 95% CI 2-sided [-0.222 to 0.040]
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 12; Test type: Superiority or Other; p = 0.8046, ANCOVA — [p-value comment as in outcome 20, analysis 1]; LS mean difference = -0.03, 95% CI 2-sided [-0.269 to 0.210]
Statistical Analysis 3: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 16; Test type: Superiority or Other; p = 0.9239, ANCOVA — [p-value comment as in outcome 20, analysis 1]; LS mean difference = 0.01, 95% CI 2-sided [-0.199 to 0.219]

21. Secondary Outcome: Change From Baseline in The Scores of DSQ Question 4 During The Treatment Period
Description: Participants' dysphagia symptoms were evaluated using the 4-item DSQ. The questionnaire was developed by the Sponsor, as an ePRO measure, according to the principles of the Final Guidance for Industry for Patient Reported Outcome Measures (PRO Guidance December 2009). All participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). Question 4 is rated as None, I had no pain (score=0), mild pain (score=1), moderate pain (score=2), severe pain (score=3), or very severe pain (score=4); 4 is the worst pain. Baseline was the DSQ score of the 14-day period before randomization. A negative change from baseline indicates that symptoms decreased.
Time Frame: Baseline, Weeks 8, 12, and 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg
Number analyzed (Participants) | 38 | 49
scores on a scale
  Week 8, n = 37, 47 | -2.52 (0.778) | -3.25 (0.690)
  Week 12, n = 36, 47 | -2.97 (0.775) | -4.89 (0.678)
  Week 16, n = 38, 47 | -3.08 (0.824) | -4.87 (0.741)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 8; Test type: Superiority or Other; p = 0.4835, ANCOVA — [p-value comment as in outcome 20, analysis 1]; LS mean difference = -0.73, 95% CI 2-sided [-2.806 to 1.339]
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 12; Test type: Superiority or Other; p = 0.0662, ANCOVA — [p-value comment as in outcome 20, analysis 1]; LS mean difference = -1.92, 95% CI 2-sided [-3.974 to 0.132]
Statistical Analysis 3: Comparison: Double-blind Placebo vs Double-blind Oral Budesonide Suspension (OBS) 2 mg; Analysis of Week 16; Test type: Superiority or Other; p = 0.1091, ANCOVA — [p-value comment as in outcome 20, analysis 1]; LS mean difference = -1.80, 95% CI 2-sided [-4.006 to 0.410]

ADVERSE EVENTS:
Description: This section reports treatment-emergent AEs (TEAEs) for the Safety Analysis Set, which was defined as all randomized participants who received at least 1 dose of double-blind study drug (placebo or OBS). Adverse events experienced during the placebo baseline period were defined as events that began before the first dose of double-blind study drug.
Groups:
- Double-blind Oral Budesonide Suspension (OBS) 2 mg: Participants took 2mg OBS (formulation MB-9) 2 mg twice daily (bid) at home for 12 weeks. Study drug was administered once in the morning after breakfast and once in the evening at bedtime; the volume per dose was 10 mL of oral liquid.
Arm/Group | Double-blind Placebo | Double-blind Oral Budesonide Suspension (OBS) 2 mg | Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg | Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/51 | 1/37 | 0/45
Other Adverse Events (participants affected / at risk) | 21/42 | 20/51 | 29/37 | 27/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=42) | Double-blind Oral Budesonide Suspension (OBS) 2 mg (N=51) | Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg (N=37) | Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg (N=45)
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=42) | Double-blind Oral Budesonide Suspension (OBS) 2 mg (N=51) | Placebo to Open-label Oral Budesonide Suspension (OBS) 2 mg (N=37) | Oral Budesonide Suspension (OBS) 2 mg to Open-label OBS 2 mg (N=45)
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 2
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 1 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 1 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 2
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 3 | 4 | 5
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 4 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 3 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.